CLINICAL TRIAL: NCT04517032
Title: ColoRectal Cancer in India: catastrOphiC expenDIture and Referral Pathways infLuencE on Presentation and Treatment
Acronym: CROCODILE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: NIHR Research Unit on Global Surgery (Unknown)
Responsible Party: Sponsor
Other Study IDs: CROC-20200503
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Cancer; Treatment Compliance; Health Care Utilization
MeSH Terms: conditions — Colorectal Neoplasms; Patient Compliance; Patient Acceptance of Health Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study to assess barriers for colorectal cancer treatment compliance in India, including quantitative assessment of catastrophic expenditure incidence and qualitative assessment of financial and non-financial barriers.

DETAILED DESCRIPTION:
Objective: To identify a vulnerable group of colorectal cancer patients in India who cannot afford or are unable to comply with a treatment plan for colorectal cancer.

Aims:

1. To identify the proportion of CRC patients suffering catastrophic expenditure due to out-of-pocket payments for cancer treatment.
2. To determine the proportion of patients who are unable to comply with the treatment plan for CRC, at 6 weeks, 3 months and 6 months after diagnosis.
3. To identify barriers and solutions to CRC treatment compliance. Design: A mixed-methods study comprising quantitative pilot data from 3 tertiary cancer centres and qualitative work from interviews with patients and healthcare professionals.

Participants: Patients diagnosed with primary colorectal cancer.

Outcomes:

Primary outcome:

• Incidence of catastrophic expenditure due to out-of-pocket payments for cancer care at 3 timepoints: 6 weeks, 3 months and 6 months after CRC diagnosis.

Secondary outcomes:

* Compliance to the initial treatment plan at three timepoints: 6 weeks, 3 months and 6 months after CRC diagnosis.
* Patients and healthcare professionals perspectives on patient compliance to CRC treatment.
* Identify the 5 main drivers (items charged to the patient) of CRC treatment cost.
* Colorectal cancer stage at the time of diagnosis.

ELIGIBILITY:
Inclusion Criteria

* Adults aged 18+ years old. AND
* Consecutive new patients with a histopathology proven colorectal cancer for whom a CRC treatment plan is made:

  * In an multi-disciplinary team meeting (MDT);
  * OR in the outpatient clinic where an MDT is not available (surgery, oncology or radiotherapy outpatient clinic).

AND

• Undergoing treatment in the hospital where the MDT took place

Exclusion Criteria

* Patients with no histopathology available
* Telephone follow-up not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive new patients with a histopathology proven colorectal cancer for whom a CRC treatment plan is made.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Catastrophic Expenditure at 6 months | 6 months after treatment decision
  Catastrophic expenditure (CE) will be defined as out of pocket payments for CRC treatment greater than 40% of patient income (assessed by an in-person questionnaire led by a researcher).

SECONDARY OUTCOMES:
Catastrophic Expenditure at 6 weeks | 6 weeks after treatment decision
  Catastrophic expenditure (CE) will be defined as out of pocket payments for CRC treatment greater than 40% of patient income (assessed by an in-person questionnaire led by a researcher).
Catastrophic Expenditure at 3 months | 3 months after treatment decision
  Catastrophic expenditure (CE) will be defined as out of pocket payments for CRC treatment greater than 40% of patient income (assessed by an in-person questionnaire led by a researcher).
Treatment compliance at 6 weeks | 6 weeks after treatment decision
  A compliant patient will be defined as undergoing or having completed the planned treatment agreed at the time of diagnosis or MDT discussion.
Treatment compliance at 3 months | 3 months after treatment decision
  A compliant patient will be defined as undergoing or having completed the planned treatment agreed at the time of diagnosis or MDT discussion.
Treatment compliance at 6 months | 6 months after treatment decision
  A compliant patient will be defined as undergoing or having completed the planned treatment agreed at the time of diagnosis or MDT discussion.
Identification of the main drivers of treatment cost | 6 months after treatment decision
  5 most expensive items or services during colorectal cancer treatment
Colorectal cancer stage at the time of diagnosis | At the time of colorectal cancer diagnosis (coincident with timing of patient enrolment in the study)
  AJCC (American Joint Committee on Cancer) guidance - 8th edition

IPD SHARING:
Plan to Share IPD: No